CLINICAL TRIAL: NCT07121283
Title: Comparison of the Difference in Bone Age Readings Among Radiologists Using Artificial Intelligence
Brief Title: Artificial Intelligence Assisted Bone Age Assessment
Status: Enrolling by invitation | Phase: Not Applicable | Type: Interventional
Sponsor: Cheng-Hsin General Hospital (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Single | Purpose: Diagnostic
Other Study IDs: (1141)113A-71
Record Dates: First submitted 2025-07-30; First posted 2025-08-13 (Actual); Last update posted 2025-08-13 (Actual); Status verified 2025-08

CONDITIONS: Bone Age

STUDY DESIGN:
Intervention Model Description: Six radiologists with different seniority (senior, intermediate, and junior) were recruited. The 200 standard films were evenly divided into two subsets: datasets A and B. A randomized crossover design with four periods (each with a 4-week duration) was arranged to minimize anticipation and carryover effects. Each radiologist who made an assessment with the aid of true AI or fake AI information could agree or disagree with the AI's predictions. The information of the fake AI was resulted from the randomization of the outputs from the true AI. Each radiologist was blinded to the existence of the fake AI.
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- True AI (Experimental)
  Interventions: Device: True AI
- Fake AI (Experimental)
  Interventions: Device: Fake AI

INTERVENTIONS:
Device: True AI — True output from bone age AI
  Arms: True AI
Device: Fake AI — Randomized output from bone age AI
  Arms: Fake AI

SUMMARY:
AI-Assisted Bone Age Assessment

DETAILED DESCRIPTION:
Artificial intelligence (AI) has gained great advancement in the application in clinical practice. However, this might introduce the automation bias, that the clinician over-rely on the incorrect advise from AI. The automation bias could have a great impact on the clinical decisions in an AI era. However, efforts to mitigate the automation bias tend to focus on upgrading AI performance and reducing bias in algorithms, which neglect the role of users. The aim of this study is to investigates the impact of the automation bias on the bone age assessment among radiologists with different seniority.

ELIGIBILITY:
Inclusion Criteria:

* Exams read by radiologists who interpret pediatric skeletal age exams and verbally consent to participate

Exclusion Criteria:

* Exams containing more than one radiograph will not be included. No further exclusion criteria will be applied on the basis of image quality metrics or manufacturers

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 8 (Estimated)
Dates: Start 2025-09-01 (Estimated); Primary Completion 2026-02-18 (Estimated); Study Completion 2026-02-18 (Estimated)

PRIMARY OUTCOMES:
Difference of Skeletal Age Estimate | Five months
  Mean absolute difference of bone age assessment between true AI-assisted and fake AI-assisted among radiologists

CONTACTS AND LOCATIONS:
Overall Officials: Yen-Huai Lin, Dr., Principal Investigator — Cheng-Hsin General Hospital
Locations (1):
- Cheng Hsin General Hospital, Taipei, Taiwan, Taiwan

IPD SHARING:
Plan to Share IPD: No